CLINICAL TRIAL: NCT03803410
Title: Comprehensive Surveillance of HCV Infecion in Uremics Under Maintenance Hemodialysis and Linking to Medical Care in Taiwan
Brief Title: Surveillance of HCV in Uremics and Linking to Medical Care
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20180325
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood test, noninvasive test for liver fibrosis — blood test of HCV serology and virology.noninvasive test including M2BPGi and fibroscan for liver fibrosis

SUMMARY:
HCV remains to prevail in the uremic patients under hemodialysis. The comprehensive surveillance in the risk population facilitates the link to care for HCV eradication.

DETAILED DESCRIPTION:
1. Taiwan has the leading prevalence and incidence of end-stage renal disease (ESRD) worldwide. Uremic patients on maintenance hemodialysis (HD) are at great risk for hepatitis C virus (HCV) infection. The prevalence and annual incidence of HCV infection in ESRD patients undergoing hemodialysis have been reported to be 10%-59% and 0.2%-6.2%, respectively.
2. HCV-related morbidities and mortality remain the major disease burden in the ESRD population. Uremic patients with HCV infection are associated with higher risk of excess risk of cardiovascular disease, hospitalization, worse quality of life, and mortality, and have more profound anemia compared to those without HCV infection..
3. Imperatively, uremic patients remain at high risk of HCV new- or re-infection in the hemodialysis units.
4. The investigators have performed a surveillance for prevalence of viral hepatitis in a collaborative group of Nephrologists and Hepatologists, the FORMOSA-LIKE group, which showed that the proportion of anti-HCV seropositivity in uremic patients is 15-19 % with the viremic rate of ~75% in Southern Taiwan in 2012. However, the update seroprevalence and disease severity of HCV infection among the uremic patients in the era of DAA in Taiwan is unknown. The current study aims to fully execute the surveillance program among the uremic population
5. Participants with HCV infection will be directly linked to medical care without gap. The concept of micro-elimination in the high risk environment would help to facilitate WHO goal of HCV elimination by 2030.
6. Understanding the potential drug-drug interaction (DDI) between directly acting antivirals (DAA) and co-medications for co-morbidities among uremic patients under maintenance hemodialysis would be helpful for decision-making when linking to care.
7. Comprehensive surveillance and link-to-care among hemodialysis units might have great impact on the improvement of both liver-related (biochemical and virological responses, and hepatic fibrosis regression) and non-liver related outcomes (monthly erythropoietin requirement and quality of life), and the transfer rate of clean zoning among HCV-viremic patients.

All uremic participants will be tested for anti-HCV antibody. HCV virology including viral loads (and genotypes if RNA seropositivity) will be further tested in patients with anti-HCV seropositivity. All infected subjects will be evaluated for the liver fibrosis by non-invasive methods including fibroscan, FIB-4 and APRI and Serum WFA(+) -M2BP. All participants with chronic hepatitis C infection will be directly referred to the collaborative Hepatology Departments in one medical center and 5 regional core hospitals for HCV treatment. The outcome of HCV-related diseases, in terms of proportion of HCV micro-elimination in HD facilities, liver-related outcomes (biochemistry improvement [ ALT and AFP decline], sustained virological response rate, and hepatic fibrosis regression) and non-liver related outcomes [monthly erythropoietin requirement, and quality of life [SF36, HCV-CLDQ] ) will be evaluated 2 years after executing link-to-care strategy.

Year 1: Universal screen, confirmative determination of HCV viremia, genotyping and disease staging, education and link-to-care for HCV treatment in FORMOSA-LIKE collaborative alliances Year 2,3: Re-evaluate liver and non-liver related outcomes, and rate of HCV clean zoning among hemodialysis units.

ELIGIBILITY:
Inclusion Criteria:

all uremic patients and medical staffs in the hemodialysis centers

Exclusion Criteria:

* patients who refuse consents

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The FORMOSA-LIKE group is a collaborative alliance of Hepatology and Nephrology in Taiwan. It contains around 2000 uremic patients with maintenance hemodialysis in 21 hemodialysis units (one medical center, 4 regional core hospitals and 16 regional clinics). The current study plan to launch a universal surveillance of HCV in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2973 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
HCV prevalence | 36 months
  To explore the current prevalence rate of hepatitis C virus (HCV) infection in uremic patients under maintenance hemodialysis in Taiwan

SECONDARY OUTCOMES:
liver fibrosis in HCV uremic patients | 36 months
  To identify the severity of liver diseases in the uremic patients under maintenance hemodialysis by transient elastography
Number of participants with potential drug-drug interaction with DAA | 36 months
  To evaluate the patient number of potential drug-drug interactions (DDI) of co-medications with DAA by checking-up through the website, https://www.hep-druginteractions.org/
Number of participants with hepatic outcome after HCV eradication | 36 months
  incidence of HCC and fibrosis regression by Fibroscan after link-to-care to antiviral therapy
Number of participants with extra-hepatic outcome after HCV eradication | 36 months
  patients with improvement of quality of life by questionnaire SF36 and HCV-CLDQ

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD.,PhD., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CF, Dai CY, Wang CW, Liang PC, Wei YJ, Tsai PC, Jang TY, Hsu PY, Jia-Jung Lee, Niu SW, Huang JC, Yeh ML, Huang CI, Hsieh MY, Lin YH, Chen SC, Chiu YW, Huang JF, Chang JM, Hwang SJ, Chuang WL, Yu ML; FORMOSA-LIKE investigators. Therapy as prevention toward HCV elimination in maintenance hemodialysis: a multi-center, prospective cohort study. Clin Kidney J. 2023 Jun 14;16(12):2429-2436. doi: 10.1093/ckj/sfad138. eCollection 2023 Dec. PMID 38046041
- [Derived] Wei YJ, Hsu PY, Lee JJ, Niu SW, Huang JC, Hsu CT, Jang TY, Yeh ML, Huang CI, Liang PC, Lin YH, Hsieh MY, Hsieh MH, Chen SC, Dai CY, Lin ZY, Chen SC, Huang JF, Chang JM, Hwang SJ, Chuang WL, Huang CF, Chiu YW, Yu ML. Evolutionary seroepidemiology of viral hepatitis and the gap in hepatitis C care cascades among uraemic patients receiving haemodialysis in Taiwan-the Formosa-Like Group. J Viral Hepat. 2021 May;28(5):719-727. doi: 10.1111/jvh.13477. Epub 2021 Feb 13. PMID 33533547
- [Derived] Yu ML, Huang CF, Wei YJ, Lin WY, Lin YH, Hsu PY, Hsu CT, Liu TW, Lee JJ, Niu SW, Huang JC, Hung TS, Yeh ML, Huang CI, Liang PC, Hsieh MY, Chen SC, Huang JF, Chang JM, Chiu YW, Dai CY, Hwang SJ, Chuang WL; FORMOSA-LIKE investigators. Establishment of an outreach, grouping healthcare system to achieve microelimination of HCV for uremic patients in haemodialysis centres (ERASE-C). Gut. 2021 Dec;70(12):2349-2358. doi: 10.1136/gutjnl-2020-323277. Epub 2020 Dec 10. PMID 33303567